CLINICAL TRIAL: NCT02644135
Title: A Pilot Study of the Safety, Tolerability, and Effectiveness of Halo to Prevent Acute Upper Respiratory Disease and Respiratory Virus Infections
Brief Title: A Pilot Study of the Safety, Tolerability, and Effectiveness of Halo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-11-33
Record Dates: First submitted 2015-12-09; First posted 2015-12-31 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Halo Oral Spray (Experimental): Based upon the preliminary studies that assessed the duration of the antimicrobial effects of Halo as reported in the preliminary studies and feasibility, subjects assigned to both study arms will be asked to spray the product intra-orally 3 times daily (Three sprays per use, total = 9 sprays per day).
  Interventions: Drug: Halo Oral Spray
- Halo Placebo (Placebo Comparator): The placebo will consist of purified sterile water without CPC - the active antiseptic. Subjects assigned to both study arms will be asked to spray the product intra-orally 3 times daily (Three sprays per use, total = 9 sprays per day).
  Interventions: Drug: Halo Placebo

INTERVENTIONS:
Drug: Halo Oral Spray — Three sprays per use, total = 9 sprays per day
  Arms: Halo Oral Spray
Drug: Halo Placebo — Three sprays per use, total = 9 sprays per day
  Arms: Halo Placebo

SUMMARY:
This is a pilot study of the safety, tolerability, and effectiveness of Halo to prevent acute upper respiratory illness and respiratory virus infections. This study will be conducted at one site (University Hospitals Case Medical Center) in healthy adults during the upcoming respiratory virus season (12/15/11 to 3/14/12). The intervention will be with Halo, a commercial product which is FDA-approved for the treatment of xerostomia. The placebo will consist of the phosphate buffered saline plus the preservatives in the Halo formulation and without CPC - the active antiseptic. This placebo was chosen as the Halo formulation without CPC serves to act as a barrier to attachment of oral pathogens, and as such is an important contributing factor to its antimicrobial activity (see above). Also, the formulation without CPC with preservatives exhibits some antibacterial and antiviral activity. Moreover, the formulation without CPC and no preservatives is easily contaminated and not practical to utilize as the placebo in these studies.

Male and female participants 18-45 years of age will be recruited and monitored for the development of, duration, and severity of clinical symptoms and signs consistent with acute respiratory disease (defined below) captured daily through diaries, and PCR confirmation of important respiratory viruses including influenza, rhinoviruses, adenoviruses, and respiratory syncytial virus during episodes of acute respiratory disease during the length of the study will be undertaken. Secondary objectives will assess the tolerance, acceptability and adherence to Halo as well as the change in the bacterial (oral streptococci and Group A streptococcus) and fungal microflora in the oropharynx. School or work absenteeism, visits to physicians' offices, emergency departments and urgent care centers will also be captured. Conventional cultures for these bacterial and fungal organisms will be pursued (see below). Throughout the study period, the safety, tolerability, acceptability and adherence to study products will be assessed.

DETAILED DESCRIPTION:
Significance and Background Respiratory tract disease is a major cause of morbidity and mortality throughout the world accounting for approximately 4 million deaths worldwide. Asthma, pneumonia, and acute bronchiolitis account for almost 22% of all pediatric hospitalizations in the United States. Pneumonia remains in the top ten causes for admission across all age groups in the United States. Much of which are directly caused by, or triggered from respiratory viruses including influenza, parainfluenza, respiratory syncytial virus (RSV), and adenovirus. In addition to these well-known pathogens, advancements in molecular and genomic techniques have increased our detection and identification of new respiratory viruses which also contribute to respiratory disease. There is also renewed attention on respiratory viruses previously considered benign, including the human rhinovirus and coronaviruses, as there is mounting evidence that these viruses can also lead to clinically severe disease. Influenza is one of the leading causes of infectious related deaths and hospitalizations in children and the 2009-10 H1N1 pandemic was especially severe in younger populations.

Respiratory disease can be caused by a variety of micro-organisms especially viruses. Despite the frequency and burden of acute respiratory infections worldwide and across all age groups, there has been limited progress in the management of treatment of respiratory virus infections aside from the use of anti-influenza drugs. The ability to prevent of acute respiratory disease has also been more limited except for the use of the influenza vaccine. The availability of a product that can be used with ease, is low cost but possesses broad spectrum antimicrobial and antiviral activity could play a major role in reducing the overall occurrence, morbidity and mortality associated with acute respiratory disease.

Moreover, upper respiratory infections are the leading cause of outpatient illness in U.S. military professionals and serve as the single greatest cause of lost workdays in the military. Unfortunately, these infections are not only prevalent, but also severe, constituting a primary cause of infectious disease hospitalization in U.S. military personnel including Navy shipboard and submarine personnel, and new recruits at basic training facilities. Military trainees and newly-mobilized troops are particularly subject to upper respiratory infection epidemic outbreaks due to their crowded living conditions, stressed working environments, and exposure to respiratory pathogens in disease-endemic areas. Additionally, the pulmonary disease resulting from ubiquitous infections are particularly impactful in high altitudes and other extreme environments common to Air Force/Navy activities.

Oasis Health Care has developed a technology and product that combines microbial barrier abilities along with a broad spectrum anti-infective agent cetylpyridinium chloride (CPC) at 0.1%. This formulation called Halo is commercially available for the over-the-counter treatment of xerostomia. The spray formulation has high mucoadhesion properties and prolonged retention time in the oral cavity. Cetylpyridinium chloride like chlorhexidine is a quarternary ammonium salt. However, due it possesses certain advantages over the latter in that it targets pathogenic bacteria while sparing beneficial ones (see below). Due to its chemical structure, CPC demonstrates significant antiviral activity especially against respiratory viruses (see below). Toxicology studies have shown no evidence of acute or chronic toxicity in animal models or irritant effect, and over-the-counter mouthwashes containing cetylpyridinium chloride have been marketed for over 45 years. Expanding the indications for the use of a cetylpyridinium-based spray formulation (Halo) as a potential formulation to prevent respiratory virus infections (cold and flu) is the long term goal. This proposal will examine the effect of Halo on the frequency and duration of clinically apparent acute respiratory infections and on respiratory virus burden as measured by PCR in young healthy adults through the respiratory virus season in Cleveland, Ohio.

Selection and enrollment of participants Study Enrollment and Withdrawal One hundred two healthy male and female participants, ages 18-45 will be enrolled in two groups. It is estimated that 204 subjects will need to be screened (2:1 screened to eligible) to enroll 102 subjects. At screening/enrollment, subjects will be stratified as to whether they received inactivated or live influenza virus vaccination. Subjects will be recruited through customary IRB-approved methods. Children, pregnant women, prisoners and other vulnerable individuals will not be enrolled.

Clinical/Laboratory Evaluations and Study Schedule Screening/Enrollment Written informed consent will be obtained before any clinical evaluations are performed. As noted in the safety section:. the study product has an acceptable safety profile and poses no significant toxicological risk to individuals. The formulation consists of ingredients with a long history of safe use in oral healthcare products.

A posterior pharyngeal and nasal swab will be obtained to ascertain baseline bacterial and fungal organisms and a multiplex PCR for respiratory viruses. Study product (after randomization) will be provided until the next scheduled visit, study procedures will be again reviewed, contact information for reaching study personnel will be provided, and study diaries will be distributed. Appointments for the 1st monthly evaluation will be made.

Scheduled Follow-up Visits At these visits, an interval medical and concomitant medication history will be obtained. Solicited and unsolicited adverse reactions will be ascertained. The study diaries will be reviewed with participants. An oropharyngeal exam will be conducted by study clinicians and a fuller symptom-directed physical exam will be performed if indicated. A posterior pharyngeal and nasal swab will be obtained at each visit to ascertain bacterial and fungal organisms and a multiplex PCR for respiratory viruses. The enrollment and interim visit pharyngeal and nasal swabs will be analysed in real time, all other swabs will be stored for future use determined by funding. Study bottles will be collected and counted. Study product will be provided until the next scheduled visit, study procedures will be again reviewed, and contact information for reaching study personnel will be revisited. Appointments for the next monthly evaluation will be made.

Final Study Visit This study visit will be conducted within 2 months after completing the last dose of Halo/Placebo. At this visit, an interval medical and concomitant medication history will be obtained. Solicited and unsolicited adverse reactions will be ascertained. An oropharyngeal exam will be conducted by study clinicians and a fuller symptom-directed physical exam will be performed if indicated.

Interim Visits Subjects will be instructed to contact study personnel in the event they develop an acute upper respiratory disease as defined above within 72 hours of onset of symptoms and signs (this allows for weekends and holidays). At these visits, an interval medical and concomitant medication history will be obtained. Solicited and unsolicited adverse reactions will be ascertained. An oropharyngeal exam will be conducted by study clinicians and a fuller symptom-directed physical exam will be performed if indicated. If pharyngitis with exudate is observed or suspected, a rapid group A streptococcal (GAS) screen will be performed. Subjects positive for Group A streptococcal infection will be given a prescription for appropriate antibiotics and a referral for follow-up care as needed. If individuals present with symptoms and signs of acute influenza fever, sore throat, myalgias, headache and chills, they will be tested for influenza and prescribed Tamiflu as needed. A posterior pharyngeal and nasal swab will be obtained to ascertain baseline bacterial and fungal organisms and a multiplex PCR for respiratory viruses. Any visit to a physician's office, emergency department, urgent care center or the need for hospitalization will be recorded. Subjects will be carefully instructed to record the duration of each symptom and sign to be recorded in the study-supplied diaries.

Statistical Analysis Sample Size Calculations Initially, primary outcomes in the control group vs. the treatment group will be compared using the t-test for independent samples, and this technique was used to estimate sample sizes. Specifically, sample size calculations were carried out assuming that the two groups will be of equal size and that the random assignment will be balanced. Further, it was assumed that an average of 2 events would occur in the control group, contrasted against an average of 1.5 events in the treated group (SD = 1), and that the average duration of illness would be 4 days and 3 days in the control and treated groups, respectively (SD = 2). Taking alpha to be 0.05, a sample size of 23 per group would allow the detection of a 25% difference in primary outcomes between the two groups with 80% power. The sample size was increased to 51 per group to account for potential losses to follow-up.

29 Randomization Based on whether the enrolled study participants have received any type of flu shot within the past 3 months, the participants will be classified as influenza vaccine recipients and non-recipients. Within each category, they will be randomly assigned to the control group or treatment group. The assignment will be balanced so that equal numbers are assigned to each group.

Interim Analysis The investigators will carry out an interim analysis when all the patients recruited have been followed for one and a half months. Since this is a pilot study, this analysis will be carried out at a stringent level of significance.

Statistical Analysis Standard techniques of descriptive statistics will be used to compare demographics and other patient characteristics in the two treatment groups. Since an additional focus of this pilot study is to obtain accurate estimates of the moments of the distributions of the outcome variables, confidence intervals will also be provided. Descriptive summaries of the number of events and duration of infection will be generated for the two groups. As stated above, the t-test will be used to compare estimates of the average number of events per person as well as the average duration of illness between the two groups. To the extent that the small sample size allows it, the investigators will utilize regression techniques for count data, using SAS GENMOD, to model the number of events per person adjusting for relevant covariates.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Ages between 18-45 years, inclusive
3. Non-tobacco/nicotine use (at least 3 months)
4. BMI of 17-35 kg/m2 inclusive
5. Able to comply with all study procedures and follow-up
6. Healthy on the basis of screening medical exam, blood chemistries, hematology, and serum pregnancy tests for females (at screening )
7. Non-pregnant or breast-feeding

Exclusion Criteria:

1. History of current use of narcotics, or recreational drug use.
2. Use of > 7 alcoholic beverages in 1 week
3. Any acute illness such as asthma, cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal (including eating disorder), endocrine/metabolic, neurologic, dermatologic, or psychiatric disease.
4. Treatment with another investigational product in the past 30 days
5. Immunocompromised status including HIV by history
6. Use of any other intra-oral product (especially antiseptic).
7. Intended use of mouthwash during study duration
8. Laboratory (screening) of creatinine > 1.5 X ULN, hemoglobin < 10.5 g/dL, platelet count ≤ 99,000/mm3, absolute neutrophil count ≤1200/ mm3, serum glucose ≥ 150 mg/dl (Subject can enroll prior to receiving lab results. Subject will be contacted if lab results are an exclusion and discontinue from study)
9. Use of any systemic antibiotic or antifungal within 30 days of screening
10. Prior or current history of seasonal allergies, chronic sinusitis or rhinitis
11. Allergy to any component of Halo
12. Oral lesions
13. Dentures
14. Dental Treatment currently in progress (implants, root canals, complex restorative procedures)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathers C, Fat DM, Boerma JT, World Health O. The global burden of disease : 2004 update. Geneva, Switzerland :: World Health Organization, 2008.
- [Background] Graham NM. The epidemiology of acute respiratory infections in children and adults: a global perspective. Epidemiol Rev. 1990;12:149-78. doi: 10.1093/oxfordjournals.epirev.a036050. PMID 2286216
- [Background] Merrill CT EA. Hospitalization in the United States, 2002. Rockville, MD: Agency for Healthcare Research and Quality. HCUP Fact Book No 6 2005; Publication number 05-0056.
- [Background] van den Hoogen BG, de Jong JC, Groen J, Kuiken T, de Groot R, Fouchier RA, Osterhaus AD. A newly discovered human pneumovirus isolated from young children with respiratory tract disease. Nat Med. 2001 Jun;7(6):719-24. doi: 10.1038/89098. PMID 11385510
- [Background] van der Hoek L, Pyrc K, Jebbink MF, Vermeulen-Oost W, Berkhout RJ, Wolthers KC, Wertheim-van Dillen PM, Kaandorp J, Spaargaren J, Berkhout B. Identification of a new human coronavirus. Nat Med. 2004 Apr;10(4):368-73. doi: 10.1038/nm1024. Epub 2004 Mar 21. PMID 15034574
- [Background] Esper F, Weibel C, Ferguson D, Landry ML, Kahn JS. Evidence of a novel human coronavirus that is associated with respiratory tract disease in infants and young children. J Infect Dis. 2005 Feb 15;191(4):492-8. doi: 10.1086/428138. Epub 2005 Jan 14. PMID 15655770
- [Background] Fouchier RA, Hartwig NG, Bestebroer TM, Niemeyer B, de Jong JC, Simon JH, Osterhaus AD. A previously undescribed coronavirus associated with respiratory disease in humans. Proc Natl Acad Sci U S A. 2004 Apr 20;101(16):6212-6. doi: 10.1073/pnas.0400762101. Epub 2004 Apr 8. PMID 15073334
- [Background] Woo PC, Lau SK, Chu CM, Chan KH, Tsoi HW, Huang Y, Wong BH, Poon RW, Cai JJ, Luk WK, Poon LL, Wong SS, Guan Y, Peiris JS, Yuen KY. Characterization and complete genome sequence of a novel coronavirus, coronavirus HKU1, from patients with pneumonia. J Virol. 2005 Jan;79(2):884-95. doi: 10.1128/JVI.79.2.884-895.2005. PMID 15613317
- [Background] Allander T, Tammi MT, Eriksson M, Bjerkner A, Tiveljung-Lindell A, Andersson B. Cloning of a human parvovirus by molecular screening of respiratory tract samples. Proc Natl Acad Sci U S A. 2005 Sep 6;102(36):12891-6. doi: 10.1073/pnas.0504666102. Epub 2005 Aug 23. PMID 16118271
- [Background] Gaynor AM, Nissen MD, Whiley DM, Mackay IM, Lambert SB, Wu G, Brennan DC, Storch GA, Sloots TP, Wang D. Identification of a novel polyomavirus from patients with acute respiratory tract infections. PLoS Pathog. 2007 May 4;3(5):e64. doi: 10.1371/journal.ppat.0030064. PMID 17480120
- [Background] Allander T, Andreasson K, Gupta S, Bjerkner A, Bogdanovic G, Persson MA, Dalianis T, Ramqvist T, Andersson B. Identification of a third human polyomavirus. J Virol. 2007 Apr;81(8):4130-6. doi: 10.1128/JVI.00028-07. Epub 2007 Feb 7. PMID 17287263
- [Background] Chua KB, Crameri G, Hyatt A, Yu M, Tompang MR, Rosli J, McEachern J, Crameri S, Kumarasamy V, Eaton BT, Wang LF. A previously unknown reovirus of bat origin is associated with an acute respiratory disease in humans. Proc Natl Acad Sci U S A. 2007 Jul 3;104(27):11424-9. doi: 10.1073/pnas.0701372104. Epub 2007 Jun 25. PMID 17592121
- [Background] Monto AS. Epidemiology of viral respiratory infections. Am J Med. 2002 Apr 22;112 Suppl 6A:4S-12S. doi: 10.1016/s0002-9343(01)01058-0. PMID 11955454
- [Background] Rakes GP, Arruda E, Ingram JM, Hoover GE, Zambrano JC, Hayden FG, Platts-Mills TA, Heymann PW. Rhinovirus and respiratory syncytial virus in wheezing children requiring emergency care. IgE and eosinophil analyses. Am J Respir Crit Care Med. 1999 Mar;159(3):785-90. doi: 10.1164/ajrccm.159.3.9801052. PMID 10051251
- [Background] Papadopoulos NG, Moustaki M, Tsolia M, Bossios A, Astra E, Prezerakou A, Gourgiotis D, Kafetzis D. Association of rhinovirus infection with increased disease severity in acute bronchiolitis. Am J Respir Crit Care Med. 2002 May 1;165(9):1285-9. doi: 10.1164/rccm.200112-118BC. PMID 11991880
- [Background] Arden KE, Nissen MD, Sloots TP, Mackay IM. New human coronavirus, HCoV-NL63, associated with severe lower respiratory tract disease in Australia. J Med Virol. 2005 Mar;75(3):455-62. doi: 10.1002/jmv.20288. PMID 15648064
- [Background] Esper F, Weibel C, Ferguson D, Landry ML, Kahn JS. Coronavirus HKU1 infection in the United States. Emerg Infect Dis. 2006 May;12(5):775-9. doi: 10.3201/eid1205.051316. PMID 16704837
- [Background] Chidekel AS, Rosen CL, Bazzy AR. Rhinovirus infection associated with serious lower respiratory illness in patients with bronchopulmonary dysplasia. Pediatr Infect Dis J. 1997 Jan;16(1):43-7. doi: 10.1097/00006454-199701000-00010. PMID 9002100
- [Background] Kim JO, Hodinka RL. Serious respiratory illness associated with rhinovirus infection in a pediatric population. Clin Diagn Virol. 1998 May 1;10(1):57-65. doi: 10.1016/s0928-0197(98)00004-x. PMID 9646002
- [Background] Malcolm E, Arruda E, Hayden FG, Kaiser L. Clinical features of patients with acute respiratory illness and rhinovirus in their bronchoalveolar lavages. J Clin Virol. 2001 Apr;21(1):9-16. doi: 10.1016/s1386-6532(00)00180-3. PMID 11255093
- [Background] Centers for Disease Control and Prevention (CDC). Surveillance for pediatric deaths associated with 2009 pandemic influenza A (H1N1) virus infection - United States, April-August 2009. MMWR Morb Mortal Wkly Rep. 2009 Sep 4;58(34):941-7. PMID 19730406
- [Background] Halasa NB. Update on the 2009 pandemic influenza A H1N1 in children. Curr Opin Pediatr. 2010 Feb;22(1):83-7. doi: 10.1097/MOP.0b013e3283350317. PMID 20068413
- [Background] Thomas TL, Garland FC, Mole D, Cohen BA, Gudewicz TM, Spiro RT, Zahm SH. Health of U.S. Navy submarine crew during periods of isolation. Aviat Space Environ Med. 2003 Mar;74(3):260-5. PMID 12650274
- [Background] Cross ER, Hermansen LA, Pugh WM, White MR, Hayes C, Hyams KC. Upper respiratory disease in deployed U.S. Navy shipboard personnel. Mil Med. 1992 Dec;157(12):649-51. PMID 1470376
- [Background] White DW, Feigley CE, McKeown RE, Hout JJ, Hebert JR. Association between barracks type and acute respiratory infection in a gender integrated Army basic combat training population. Mil Med. 2011 Aug;176(8):909-14. doi: 10.7205/milmed-d-10-00418. PMID 21882781
- [Background] Sanchez JL, Binn LN, Innis BL, Reynolds RD, Lee T, Mitchell-Raymundo F, Craig SC, Marquez JP, Shepherd GA, Polyak CS, Conolly J, Kohlhase KF. Epidemic of adenovirus-induced respiratory illness among US military recruits: epidemiologic and immunologic risk factors in healthy, young adults. J Med Virol. 2001 Dec;65(4):710-8. doi: 10.1002/jmv.2095. PMID 11745936
- [Background] Zhanel GG, Kirkpatrick ID, Hoban DJ, Kabani AM, Karlowsky JA. Influence of human serum on pharmacodynamic properties of an investigational glycopeptide, LY333328, and comparator agents against Staphylococcus aureus. Antimicrob Agents Chemother. 1998 Sep;42(9):2427-30. doi: 10.1128/AAC.42.9.2427. PMID 9736576
- [Background] Zhanel GG, Saunders DG, Hoban DJ, Karlowsky JA. Influence of human serum on antifungal pharmacodynamics with Candida albicans. Antimicrob Agents Chemother. 2001 Jul;45(7):2018-22. doi: 10.1128/AAC.45.7.2018-2022.2001. PMID 11408217
- [Background] Manavathu EK, Ramesh MS, Baskaran I, Ganesan LT, Chandrasekar PH. A comparative study of the post-antifungal effect (PAFE) of amphotericin B, triazoles and echinocandins on Aspergillus fumigatus and Candida albicans. J Antimicrob Chemother. 2004 Feb;53(2):386-9. doi: 10.1093/jac/dkh066. Epub 2004 Jan 16. PMID 14729762
- [Background] Clancy CJ, Huang H, Cheng S, Derendorf H, Nguyen MH. Characterizing the effects of caspofungin on Candida albicans, Candida parapsilosis, and Candida glabrata isolates by simultaneous time-kill and postantifungal-effect experiments. Antimicrob Agents Chemother. 2006 Jul;50(7):2569-72. doi: 10.1128/AAC.00291-06. PMID 16801448
- [Background] Chandra J, Mukherjee PK, Ghannoum MA. In vitro growth and analysis of Candida biofilms. Nat Protoc. 2008;3(12):1909-24. doi: 10.1038/nprot.2008.192. PMID 19180075
- [Background] Mukherjee PK, Chandra J, Jurevic RJ, Ghannoum A, Ghannoum MA. Activity of Oasis™ and Biotene™ mouthwashes against microbial biofilmsIADR/AADR/CADR 89th General Session. San Diego, CA: IADR/AADR, 2011.
- [Background] Rouabhia M, Deslauriers N. Production and characterization of an in vitro engineered human oral mucosa. Biochem Cell Biol. 2002;80(2):189-95. doi: 10.1139/o01-237. PMID 11989714
- [Background] Mukherjee PK, Mohamed S, Chandra J, Kuhn D, Liu S, Antar OS, Munyon R, Mitchell AP, Andes D, Chance MR, Rouabhia M, Ghannoum MA. Alcohol dehydrogenase restricts the ability of the pathogen Candida albicans to form a biofilm on catheter surfaces through an ethanol-based mechanism. Infect Immun. 2006 Jul;74(7):3804-16. doi: 10.1128/IAI.00161-06. PMID 16790752
- [Background] Brittain-Long R, Nord S, Olofsson S, Westin J, Anderson LM, Lindh M. Multiplex real-time PCR for detection of respiratory tract infections. J Clin Virol. 2008 Jan;41(1):53-6. doi: 10.1016/j.jcv.2007.10.029. PMID 18093871
- [Background] Mourez T, Bergeron A, Ribaud P, Scieux C, de Latour RP, Tazi A, Socie G, Simon F, LeGoff J. Polyomaviruses KI and WU in immunocompromised patients with respiratory disease. Emerg Infect Dis. 2009 Jan;15(1):107-9. doi: 10.3201/eid1501.080758. PMID 19116066
- [Background] Chow BD, Esper FP. The human bocaviruses: a review and discussion of their role in infection. Clin Lab Med. 2009 Dec;29(4):695-713. doi: 10.1016/j.cll.2009.07.010. PMID 19892229
- [Derived] Mukherjee PK, Esper F, Buchheit K, Arters K, Adkins I, Ghannoum MA, Salata RA. Randomized, double-blind, placebo-controlled clinical trial to assess the safety and effectiveness of a novel dual-action oral topical formulation against upper respiratory infections. BMC Infect Dis. 2017 Jan 14;17(1):74. doi: 10.1186/s12879-016-2177-8. PMID 28088167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Halo Oral Spray | Halo Placebo
Started | 50 | 44
Completed | 50 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Halo Oral Spray | Halo Placebo | Total
Number analyzed (Participants) | 50 | 44 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 44 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.14 (6.73) | 24.86 (6.47) | 24.86 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Develop Acute Respiratory Illnesses When Using Halo vs Placebo
Time Frame: Through study duration, an average of 3 months
Population: Among the 94 enrolled individuals, there were six participants who presented to the clinic for clinical confirmation and collection of oral and nasal swabs related to the development of URIs symptoms (Confirmed URIs Episode).
Measure: Number; unit: participants
Arm/Group | Halo Oral Spray | Halo Placebo
Number analyzed (Participants) | 50 | 44
participants | 2 | 4

2. Secondary Outcome: Number of Acute Respiratory Illnesses
Description: Measured by medical record review.
Time Frame: Through study duration, an average of 3 months
Measure: Number; unit: Number of acute respiratory illnesses
Arm/Group | Halo Oral Spray | Halo Placebo
Number analyzed (Participants) | 50 | 44
Number of acute respiratory illnesses | 4 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Halo Oral Spray | Halo Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/44
Other Adverse Events (participants affected / at risk) | 4/50 | 5/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Halo Oral Spray (N=50) | Halo Placebo (N=44)
headache (General disorders) | 2 (2) | 2 (2)
Anxiety (General disorders) | 1 (1) | 1 (1)
Labial mucosal injury (General disorders) | 0 | 1 (1)
Muscle strain (General disorders) | 0 (0) | 1 (1)
extremity rash (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No